CLINICAL TRIAL: NCT07240246
Title: Effect of a Dietary Supplement (FitLine TopShape) on the Incretin Response
Brief Title: Effect of a Dietary Supplement on Hormones Involved in Appetite Regulation in Overweight and Obese Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FFoQSI - Austrian Competence Centre for Feed and Food Quality, Safety & Innovation (Other)
Collaborators: Salzburger Universitätsklinkum (Unknown); University of Applied Sciences Upper Austria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1098/2025
Record Dates: First submitted 2025-09-24; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: GLP-1; Obesity &Amp; Overweight; Dietary Supplement
Keywords: Obesity; Overweight; Incretins; Dietary Supplement; Plant Extract; Appetite Regulation; Dipeptidyl-Peptidase IV; Glucagon-Like Peptide 1; Gastric Inhibitory Polypeptide
MeSH Terms: conditions — Obesity; Overweight | interventions — Plant Extracts

STUDY DESIGN:
Intervention Model Description: The study is designed as a 3-month parallel, double-blind, randomised, placebo-controlled trial involving adults who are overweight or obese (BMI 25-40; age 18-50 years). Participants will be randomised in a 1:1 ratio to two arms: (1) placebo and (2) intervention group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Supplement (Active Comparator): Participants receive a dietary supplement: Capsule preparation containing hypromellose, calcium phosphate, inulin, yeast extract (Saccharomyces cerevisiae), bitter melon extract, green coffee bean extract, white mulberry extract, purslane extract, peppermint leaf extract, dandelion extract, green mate extract, zinc gluconate, ginger extract, biotin and yellow iron oxide (E172 - capsule colouring)
  Interventions: Dietary Supplement: Intervention: Dietary Supplement with Plant Extracts
- Placebo (Placebo Comparator): Participants receive a capsule preparation containing hypromellose, calcium phosphate, inulin and yellow iron oxide (E172 - capsule colouring agent)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Intervention: Dietary Supplement with Plant Extracts — Capsule containing a blend of plant extracts, administered twice daily three capsules (total six capsules), 30-60 minutes before main meals, for 12 weeks.
  Arms: Dietary Supplement
Other: Placebo — Matching capsule without active plant extracts, administered twice daily three capsules (in total six), 30-60 minutes before main meals, for 12 weeks.
  Arms: Placebo

SUMMARY:
Obesity is a chronic condition linked to numerous health risks and affects more than one billion people worldwide. While pharmacological treatments such as incretin-based therapies are available, they may have side effects, are not suitable for all patients, and adherence can be limited. Dietary supplements that influence appetite and satiety may represent an alternative or complementary approach.

This study will evaluate whether a dietary supplement containing plant extracts stimulates the intestinal incretin response. The primary focus is the effect on glucagon-like peptide-1 (GLP-1) secretion. Secondary outcomes include dipeptidyl peptidase-4 (DPP-4), gastric inhibitory peptide (GIP), and insulin, as well as measures of appetite, satiety, food intake, and anthropometrics.

The trial is designed as a 12-week, double-blind, randomized, placebo-controlled parallel-group study in adults with overweight or obesity (BMI 25-40, age 18-50). Participants will receive either the dietary supplement or placebo. Blood samples will be collected at baseline and after 12 weeks, both fasting and following capsule intake and a standardized liquid meal. Anthropometric measurements and visual analog scales (VAS) for hunger and satiety will also be assessed.

DETAILED DESCRIPTION:
Obesity is a chronic disease associated with a wide range of adverse health outcomes, including type 2 diabetes mellitus, coronary heart disease, and other metabolic disorders. The global rise in obesity is driven in part by sedentary lifestyles and the widespread availability of calorie-dense foods. According to the World Health Organization, over one billion people worldwide are affected by obesity (BMI ≥ 30 kg/m²), with even more classified as overweight (BMI ≥ 25 kg/m²). This trend poses significant challenges not only to individual health but also to public health systems due to the high costs of treating obesity-related complications.

Lifestyle modification remains the cornerstone of effective weight management. For individuals with overweight but without comorbidities, the primary goal is to prevent further weight gain through increased physical activity and dietary adjustments. Evidence suggests that even modest weight loss of 5-10% can lead to clinically meaningful improvements in cardiovascular risk factors.

In this context, dietary supplements that support appetite regulation and satiety enhancement are of growing interest. Several plant extracts-including bitter melon, yerba mate, green tea, turmeric, and others-have shown potential to stimulate the secretion of glucagon-like peptide-1 (GLP-1), a gut hormone involved in satiety signaling, appetite suppression, and insulin secretion.

GLP-1 is secreted by intestinal L-cells in response to food intake and acts via GLP-1 receptors. However, native GLP-1 has a short half-life of approximately two minutes due to rapid degradation by the enzyme dipeptidyl peptidase-4 (DPP-4). Therefore, strategies that stimulate GLP-1 secretion or inhibit DPP-4 activity may enhance satiety and support weight control. While promising, current evidence is largely limited to in vitro and animal studies, and human data are lacking.

This randomized, double-blind, placebo-controlled clinical trial aims to investigate the effects of a commercially available dietary supplement (FitLine TopShape) on GLP-1 secretion and related metabolic parameters. The supplement contains extracts from purslane, bitter melon, dandelion, mulberry, yerba mate, and green coffee beans. Preliminary user data from an observational study (n=40) suggest that daily intake of the supplement may increase satiety and promote weight loss (mean reduction: -1.32 kg over four weeks; unpublished). In vitro assays indicate that the bioactive compounds may reduce DPP-4 activity and increase GLP-1 secretion (unpublished).

The primary objective of this study is to assess the effect of the supplement on GLP-1 secretion. Secondary outcomes include changes in DPP-4 activity, gastric inhibitory peptide (GIP), insulin, and C-peptide levels. Subjective measures of satiety, appetite, and food intake will be collected via validated questionnaires. Anthropometric data (weight, height, waist and hip circumference) will be recorded at baseline and after 12 weeks of intervention.

Participants (BMI 25-40 kg/m², age 18-50 years) will be randomized 1:1 to receive either the dietary supplement or placebo for 12 weeks. Blood samples will be collected in fasting state and at multiple time points post-ingestion of the capsule and a standardized liquid meal. The study will evaluate both acute hormonal responses and long-term effects on weight control.

ELIGIBILITY:
Inclusion Criteria:

* Signing the consent form
* BMI 25-40 kg/m²
* Age 18-50 years

Exclusion Criteria:

* Known allergy to ingredients in the administered substances
* Type 1 or 2 diabetes
* Pregnancy
* Breastfeeding mothers
* Acute infectious disease
* Renal insufficiency

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
GLP-1 secretion | 12 weeks
  Taking the dietary supplement over a period of 12 weeks changes GLP-1 secretion (area under the curve (AUC) over 60 minutes) in overweight or obese subjects* compared to the start of the study (AUC over 60 minutes).

SECONDARY OUTCOMES:
Intervention vs. Placebo | 12 weeks
  Taking the dietary supplement over a period of 12 weeks changes GLP-1, DPP-4, GIP, and insulin secretion (AUC over 60 min) in overweight or obese subjects* compared to taking a placebo (AUC over 60 min).
Liquid Meal | 12 weeks
  Taking the dietary supplement over a period of 12 weeks changes GLP-1, DPP-4, GIP, and insulin secretion (AUC over 60 min) in overweight or obese subjects* after consuming a standardised liquid meal compared to intake at the start of the study (AUC over 60 min).
Liquid Meal: Intervention vs. Placebo | 12 weeks
  Taking the dietary supplement over a period of 12 weeks changes GLP-1, DPP-4, GIP, and insulin secretion (AUC over 60 min) in overweight or obese subjects* after consuming a standardised liquid meal compared to taking a placebo (AUC over 60 min).
Body weight | 12 weeks
  Taking the dietary supplement over a period of 12 weeks leads to changes in body weight (kg).
Body mass index (BMI) in kg/m² | 12 weeks
  BMI in kg/m² will be determined using weight (kg) and height (m). Taking the dietary supplement over a period of 12 weeks leads to changes in BMI.
Abdominal Circumference | 12 weeks
  Taking the dietary supplement over a period of 12 weeks leads to changes in the abdominal circumference (cm).
Waist to Hip Ratio | 12 weeks
  Taking the dietary supplement leads to changes in the waist-hip ratio (cm waist/cm hip = WHR).
Changes in Control of Eating Questionnaire (CoEQ) | 12 weeks
  Participants report on their control of eating by answering the Control of Eating Questionnaire (CoEQ) with 19 questions. Rating on a horizontal, non-calibrated line of 10 cm, ranging from very low (0) to very high (10).
Visual analog scale (VAS) to assess hunger | 12 weeks
  Visual analog scale (VAS) to assess hunger on a horizontal, non-calibrated line of 10 cm, ranging from not hungry at all (0) to very hungry (10)
Visual analog scale (VAS) to assess satiation | 12 weeks
  Visual analog scale (VAS) to assess satiation (process that leads to the termination of eating) on a horizontal, non-calibrated line of 10 cm, ranging from completely empty (0) to cannot eat another bite (10)
Visual analog scale (VAS) to assess desire to eat | 12 weeks
  Visual analog scale to assess desire to eat on a horizontal, non-calibrated line of 10 cm, ranging from very low (0) to very strong (10)
Visual analog scale (VAS) to assess the amount that can be eaten right now | 12 weeks
  Visual analog scale to assess the amount that can be eaten right now on a horizontal, non-calibrated line of 10 cm, ranging from not at all (0) to a large amount (10)
Visual analog scale (VAS) to assess satiety | 12 weeks
  Visual analog scale to assess satiety (feeling of fullness that persists after eating suppressing further energy intake) on a horizontal, non-calibrated line of 10 cm, ranging from not full at all (0) to totally full (10)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weghuber, Prim. Univ. Prof. Dr., Study Director — Salzburger Universitätsklinikum
Locations (1):
- Salzburger Universitätsklinikum, Salzburg, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu CY, Huang CJ, Huang LH, Chen IJ, Chiu JP, Hsu CH. Effects of green tea extract on insulin resistance and glucagon-like peptide 1 in patients with type 2 diabetes and lipid abnormalities: a randomized, double-blinded, and placebo-controlled trial. PLoS One. 2014 Mar 10;9(3):e91163. doi: 10.1371/journal.pone.0091163. eCollection 2014. PMID 24614112
- [Background] Stenlid R, Manell H, Halldin M, Kullberg J, Ahlstrom H, Manukyan L, Weghuber D, Paulmichl K, Zsoldos F, Bergsten P, Forslund A. High DPP-4 Concentrations in Adolescents Are Associated With Low Intact GLP-1. J Clin Endocrinol Metab. 2018 Aug 1;103(8):2958-2966. doi: 10.1210/jc.2018-00194. PMID 29850829
- [Background] Stenlid R, Cerenius SY, Wen Q, Aydin BK, Manell H, Chowdhury A, Kristinsson H, Ciba I, Gjessing ES, Morwald K, Gomahr J, Heu V, Weghuber D, Forslund A, Bergsten P. Adolescents with obesity treated with exenatide maintain endogenous GLP-1, reduce DPP-4, and improve glycemic control. Front Endocrinol (Lausanne). 2023 Nov 1;14:1293093. doi: 10.3389/fendo.2023.1293093. eCollection 2023. PMID 38027106
- [Background] Dalton M, Finlayson G, Hill A, Blundell J. Preliminary validation and principal components analysis of the Control of Eating Questionnaire (CoEQ) for the experience of food craving. Eur J Clin Nutr. 2015 Dec;69(12):1313-7. doi: 10.1038/ejcn.2015.57. Epub 2015 Apr 8. PMID 25852028
- [Background] Gabe MBN, Breitschaft A, Knop FK, Hansen MR, Kirkeby K, Rathor N, Adrian CL. Effect of oral semaglutide on energy intake, appetite, control of eating and gastric emptying in adults living with obesity: A randomized controlled trial. Diabetes Obes Metab. 2024 Oct;26(10):4480-4489. doi: 10.1111/dom.15802. Epub 2024 Jul 31. PMID 39082206
- [Background] Muller TD, Finan B, Bloom SR, D'Alessio D, Drucker DJ, Flatt PR, Fritsche A, Gribble F, Grill HJ, Habener JF, Holst JJ, Langhans W, Meier JJ, Nauck MA, Perez-Tilve D, Pocai A, Reimann F, Sandoval DA, Schwartz TW, Seeley RJ, Stemmer K, Tang-Christensen M, Woods SC, DiMarchi RD, Tschop MH. Glucagon-like peptide 1 (GLP-1). Mol Metab. 2019 Dec;30:72-130. doi: 10.1016/j.molmet.2019.09.010. Epub 2019 Sep 30. PMID 31767182
- [Background] Smith NK, Hackett TA, Galli A, Flynn CR. GLP-1: Molecular mechanisms and outcomes of a complex signaling system. Neurochem Int. 2019 Sep;128:94-105. doi: 10.1016/j.neuint.2019.04.010. Epub 2019 Apr 17. PMID 31002893
- [Background] Adam TC, Westerterp-Plantenga MS. Glucagon-like peptide-1 release and satiety after a nutrient challenge in normal-weight and obese subjects. Br J Nutr. 2005 Jun;93(6):845-51. doi: 10.1079/bjn20041335. PMID 16022753
- [Background] Yumuk V, Tsigos C, Fried M, Schindler K, Busetto L, Micic D, Toplak H; Obesity Management Task Force of the European Association for the Study of Obesity. European Guidelines for Obesity Management in Adults. Obes Facts. 2015;8(6):402-24. doi: 10.1159/000442721. Epub 2015 Dec 5. PMID 26641646
- [Background] Aaseth J, Ellefsen S, Alehagen U, Sundfor TM, Alexander J. Diets and drugs for weight loss and health in obesity - An update. Biomed Pharmacother. 2021 Aug;140:111789. doi: 10.1016/j.biopha.2021.111789. Epub 2021 May 31. PMID 34082399
- [Background] Ackermann RT, Edelstein SL, Narayan KM, Zhang P, Engelgau MM, Herman WH, Marrero DG; Diabetes Prevention Program Research Group. Changes in health state utilities with changes in body mass in the Diabetes Prevention Program. Obesity (Silver Spring). 2009 Dec;17(12):2176-81. doi: 10.1038/oby.2009.114. Epub 2009 Apr 23. PMID 19390518
- [Background] Planes-Munoz D , Lopez-Nicolas R , Gonzalez-Bermudez CA , Ros-Berruezo G , Frontela-Saseta C . In vitro effect of green tea and turmeric extracts on GLP-1 and CCK secretion: the effect of gastrointestinal digestion. Food Funct. 2018 Oct 17;9(10):5245-5250. doi: 10.1039/c8fo01334a. PMID 30226521
- [Background] Cooper-Leavitt ET, Shin MJ, Beus CG, Chiu AT, Parker G, Radford JH, Evans EP, Edwards IT, Arroyo JA, Reynolds PR, Bikman BT. The Incretin Effect of Yerba Mate (Ilex paraguariensis) Is Partially Dependent on Gut-Mediated Metabolism of Ferulic Acid. Nutrients. 2025 Feb 9;17(4):625. doi: 10.3390/nu17040625. PMID 40004954
- [Background] Romdhoni MF, Doewes M, Soetrisno S, Febrinasari RP. Antidiabetic Activity of Momordica charantia Extracts Through Incretin Pathway in Streptozotocin-Nicotinamide Induced Diabetic Rat Depends on Dose Differences. Avicenna J Med Biotechnol. 2025 Jan-Mar;17(1):47-55. doi: 10.18502/ajmb.v17i1.17677. PMID 40094091
- [Background] Bhat GA, Khan HA, Alhomida AS, Sharma P, Singh R, Paray BA. GLP-I secretion in healthy and diabetic Wistar rats in response to aqueous extract of Momordica charantia. BMC Complement Altern Med. 2018 May 18;18(1):162. doi: 10.1186/s12906-018-2227-4. PMID 29776414
- [Background] Gleason PP, Urick BY, Marshall LZ, Friedlander N, Qiu Y, Leslie RS. Real-world persistence and adherence to glucagon-like peptide-1 receptor agonists among obese commercially insured adults without diabetes. J Manag Care Spec Pharm. 2024 Aug;30(8):860-867. doi: 10.18553/jmcp.2024.23332. Epub 2024 May 8. PMID 38717042
- [Background] Melson E, Ashraf U, Papamargaritis D, Davies MJ. What is the pipeline for future medications for obesity? Int J Obes (Lond). 2025 Mar;49(3):433-451. doi: 10.1038/s41366-024-01473-y. Epub 2024 Feb 1. PMID 38302593
- [Background] World health statistics 2024: monitoring health for the SDGs, Sustainable Development Goals. Geneva: World Health Organization; 2024. Licence: CC BY-NC-SA 3.0 IGO.